CLINICAL TRIAL: NCT03270982
Title: Comprehensive Segmental Revision System
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.GE5
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Disease; Oncology; Revision Surgery; Trauma; Rheumatoid Arthritis
Keywords: Non Inflammatory Degenerative Joint Disease; Rheumatoid Arthritis; Revision where other devices have failed; Correction of functional deformity; Oncology Applications; Treatment of acute or Chronic fractures
MeSH Terms: conditions — Neoplasms; Wounds and Injuries; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Comprehensive SRS Replacement: Comprehensive SRS Device
  Interventions: Device: Comprehensive SRS Replacement

INTERVENTIONS:
Device: Comprehensive SRS Replacement — This system consist of a proximal humeral replacement, distal humeral replacement, or total humeral replacement.

SUMMARY:
Clinical Data evaluation to document the performance and clinical outcomes of the Comprehensive Segmental Revision System.

DETAILED DESCRIPTION:
The Purpose of this multi centre clinical data evaluation is to document the performance and clinical outcomes of the Comprehensive Segmental revision System. The data gathered will be collated and used to provide feedback to designing engineers, support marketing efforts, answer potential questions from reimbursement agencies, and will serve as part of Zimmer Biomets Post Market Surveillance.

The Comprehensive Segmental Revision System consists of a proximal humeral replacement system (shoulder prosthesis), a distal humeral replacement system (elbow prosthesis) and of a total humeral replacement system (shoulder and elbow prosthesis connected by a humeral coupler).

Patient outcomes will be measured by using measurement tools that have been extensively used and referred to in the literature. Specifically, the quickDASH will be used for all cases enrolled in the study. In addition, the Constant and Murley Score may be used for shoulder applications, the Liverpool Elbow Score may be used for elbow applications and the MSTS Score may be used for tumor cases.

The study population will be compromised of males and females that are eligible according to the inclusion/exclusion criteria. The study will last for at least ten (10) years from the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Non Inflammatory Degenerative joint disease, including osteoarthritis, and avascular necrosis
* Rheumatoid arthritis
* Revision where other devices or treatments have failed
* Correction of functional deformity
* Oncology applications including bone loss due to tumour resection

Exclusion Criteria:

* Sepsis ( active)
* Infection ( active)
* Osteomyelitis (active)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will come from Primary Care Clinics
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Implant survivorship assessed according to the implant revisions | 10 years
  Implant survivorship assessed counting the number of implant revisions

SECONDARY OUTCOMES:
Clinical patient outcome measure: QuickDASH | Pre-operative and at 6 months, 1 year, 3 years and 5 years post-operative
  The QuickDASH score will be used to measure physical function and symptoms of the upper limb in patients to be treated/treated with the Comprehensive SRS products.
Clinical patient outcome measure: Constant-Murley Score | Pre-operative and at 6 months, 1 year, 3 years and 5 years post-operative
  The Constant-Murley score may be used to define the level of pain and the ability to carry out the normal daily activities in patients to be treated/treated with the Comprehensive SRS products. The score consists of objective (ROM, strength) and subjective (pain, functional assessment) variables.
Clinical patient outcome measure: Liverpool Elbow Score | Pre-operative and at 6 months, 1 year, 3 years and 5 years post-operative
  The Liverpool Elbow Score may be used to define elbow condition, function and pain in patients to be treated/treated with the Comprehensive SRS products.The score consists of two components: one patient-rated part and another part that can be measured objectively.
Clinical patient outcome measure: Musculoskeletal Tumour Society Scoring System (MSTS) | 6 months, 1 year, 3 years and 5 years post-operative
  The MSTS Score may be used as a functional measure for patients with sarcoma involving the upper limb. The score includes 6 measures (pain, function, emotional acceptance, hand position, manual dexterity, lifting ability) each measure with a maximum of 5 points. The maximum overall score is 30 points. The score is designed to be used after the procedure and is therefore only collected post-operatively.
Safety is assessed according to the number of complications | 10 years
  Safety is assessed according to the number of complications which are collected via adverse event forms

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, Study Director — Clinical Operations Director Zimmer Biomet EMEA
Locations (4):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada
- Department of Orthopedic Surgery, Rigshospitalet University of Copenhagen, Copenhagen, Denmark
- United Kingdom (2):
  - Royal Gwent Hospital, Newport, Wales
  - Royal Liverpool University Hospital, Liverpool